CLINICAL TRIAL: NCT04035655
Title: Sub-study of the NEURODOC Project (Electrophysiological Evaluation of Consciousness in Patients With Disorders of Consciousness During Standard Care Procedures): Neurophysiological Evaluation of a Routine Care Open Label tDCS Session
Brief Title: Sub-study of the NEURODOC Project : Neurophysiological Evaluation of a Routine Care Open Label tDCS Session
Acronym: Neurodoc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, LIONEL NACCACHE, Professor, Groupe Hospitalier Pitie-Salpetriere
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A01385-40
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Disorder of Consciousness; Traumatic Brain Injury; Anoxic Brain Injury; Stroke
Keywords: Disorders of consciousness; Transcranial direct current stimulation; Electroencephalography; Electrophysiological signatures of consciousness; Coma Recovery Scale - Revised
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries, Traumatic; Hypoxia-Ischemia, Brain; Stroke | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Electrophysiological evaluation of a routine care intervention: single session of left dorso-lateral transcranial direct current stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Clinical and electrophysiological evaluation of tDCS session (Experimental): In this prospective case-control study, the investigator's main goal was to evaluate the impact of a single standard-care tDCS session on brain activity (EEG).
  The effect of a single 20 minutes 2 mA tDCS session with the anode placed over the left dorsolateral prefrontal cortex and the cathode over the right supraorbital cortex administered as routine care were evaluated by combined behavioral and electrophysiological assessments immediately before and after the stimulation.
  The study consisted of the following interventions, administered immediately before and after the stimulation session:
  * detailed behavioral assessment by the Coma Recovery Scale-Revised (CRS-R)
  * 5 minutes resting state high-density EEG recordings and 6 minutes auditory oddball paradigm immediately.
  Additionally, clinical anatomical MRI (T1) acquired as routine care were used to model the estimated tDCS-induced electric fields in the entire head of patients, based on available T1-weighted MRI.
  Interventions: Behavioral: Coma Recovery Scale - revised; Diagnostic Test: Electrophysiological recordings

INTERVENTIONS:
Behavioral: Coma Recovery Scale - revised — Assessment of the level of consciousness by the dedicated Coma Recovery Scale - Revised, current gold-standard in consciousness level assessment.
  Assessment before and after the tDCS session (immediately before and after the electrophysiological assessment, see below).
  Other Names: CRS-R
Diagnostic Test: Electrophysiological recordings — The electrophysiological assessment consisted of:
  * a 5 minutes resting state high-density EEG recording
  * a approximately 6 minutes auditory oddball paradigm These two procedures were administered immediately before and after the tDCS session
  Other Names: EEG

SUMMARY:
Limited treatments are available to improve consciousness in severely brain injured patients. Transcranial Direct Current stimulation (tDCS) is one of the few therapeutics that showed evidence of efficacy to increase level of consciousness and functional communication in some Minimally Conscious State (MCS) patients, and in some Vegetative State (VS) patients.

However the mechanisms by which tDCS improves consciousness are poorly understood and the electrophysiological effects of such a stimulation have never been studied in disorders of consciousness patients.

In this study, the investigators will use detailed clinical examinations and electrophysiological assessments (quantitative high-density EEG and event-related potentials) to assess the effect of a open-label single session of left dorsolateral prefrontal cortex tDCS stimulation administered as routine care.

DETAILED DESCRIPTION:
Limited treatments are available to improve consciousness in severely brain injured patients. Transcranial Direct Current stimulation (tDCS) is one of the few therapeutics that showed evidence of efficacy to increase level of consciousness and functional communication in some Minimally Conscious State (MCS) patients, and in some Vegetative State (VS) patients (1, 2, 3, 4), with no side effects reported.

However the mechanisms by which tDCS improves consciousness are poorly understood and the electrophysiological effects of the stimulation have never been studied in disorders of consciousness patients.

In this study, the investigators will use detailed clinical examinations (Coma Recovery Scale - Revised (5)) and electrophysiological assessments (quantitative high-density EEG and event-related potentials) (6, 7) and event-related potentials (8, 9) together with a standard morphological MRI to assess the effect of a open-label single session of left dorsolateral prefrontal cortex tDCS stimulation administered as routine care.

The primary goal is to investigate electrophysiological response to tDCS and its relation to behavioral response to better understand how tDCS affects consciousness in disorders of consciousness patients.

References:

1. Angelakis, E. et al. Transcranial Direct Current Stimulation Effects in Disorders of Consciousness. Arch. Phys. Med. Rehabil. 95, 283-289 (2014).
2. Thibaut, A., Bruno, M.-A., Ledoux, D., Demertzi, A. & Laureys, S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology 82, 1112-1118 (2014).
3. Thibaut, A. et al. Controlled clinical trial of repeated prefrontal tDCS in patients with chronic minimally conscious state. Brain Inj. 1-9 (2017). doi:10.1080/02699052.2016.1274776
4. Martens, G. et al. Randomized controlled trial of home-based 4-week tDCS in chronic minimally conscious state. Brain Stimulat. (2018). doi:10.1016/j.brs.2018.04.021
5. Giacino, J. T. & Kalmar, K. Diagnostic and prognostic guidelines for the vegetative and minimally conscious states. Neuropsychol. Rehabil. 15, 166-174 (2005).
6. Sitt, J. D. et al. Large scale screening of neural signatures of consciousness in patients in a vegetative or minimally conscious state. Brain 137, 2258-2270 (2014).
7. Engemann, D. A. et al. Robust EEG-based cross-site and cross-protocol classification of states of consciousness. Brain J. Neurol. 141, 3179-3192 (2018).
8. Bekinschtein, T. A. et al. Neural signature of the conscious processing of auditory regularities. Proc. Natl. Acad. Sci. 106, 1672-1677 (2009).
9. Faugeras, F. et al. Event related potentials elicited by violations of auditory regularities in patients with impaired consciousness. Neuropsychologia 50, 403-418 (2012).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Disorder of consciousness assessed by CRS-R (VS, MCS, exitMCS)
* Patients with stable clinical examination (even in intensive care unit)
* Structural brain injury confirmed by cerebral imaging (MRI or TDM)

Exclusion Criteria:

* Refractory status epilepticus
* Known preexisting severe neurodegenerative disease (ie: Alzheimer disease, Lewy body dementia, ...)
* MRI contraindication: metallic intra-cranial implants, pacemaker or implantable cardioverter-defibrillator, cranial prosthesis
* Pregnant, parturient or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Support vector machine multivariate prediction of consciousness from resting state EEG markers | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change from baseline of the predicted probability of conscious state, ie. to be classified a in a 'minimally conscious state' as opposed to be classified as in a 'vegetative state'.
  The prediction will be based on a set of markers extracted from the EEG (power spectra, information theory, complexity and connectivity markers) and will use a support vector machine classifier algorithm train on a validated database. See Sitt et al., Brain et al. 2014. for details on the EEG preprocessing, markers extraction, support vector machine algorithm and training database.
Evoked response potential during auditory oddball paradigm | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change of the Evoked Response Potentials recorded during the auditory oddball paradigm

SECONDARY OUTCOMES:
Resting state EEG individual markers | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  In addition to the multivariate classification from the EEG, the response to stimulation will be evaluated on several quantitative markers derived from the EEG: power spectrum, complexity and connectivity assessed by the weighted symbolic mutual information (King & Sitt, Current Biology 2013; Sitt, Brain 2014; Engemann & Raimondo, Brain 2018)
State of consciousness | Two time points: immediately before (baseline) and immediately after stimulation (post-stimulation)
  Change of the Coma Recovery Scale-Revised scores (CRS-R, Giacino et al. Neurology 2002 and Kalmar et al., Neuropsychol Rehabil 2005) between before and after stimulation (CRS-R post stimulation - CRS-R before stimulation). The CRS-R score is a qualitative and quantitative scales ranking predefined behaviors elicited by the patients in the following six subscales, auditory function, visual function, motor function, verbal and oromotor function, communication and wakefulness, the sum of which give a total score ranging from 0 to 23. Higher values of the scale mean a better state of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Naccache, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angelakis E, Liouta E, Andreadis N, Korfias S, Ktonas P, Stranjalis G, Sakas DE. Transcranial direct current stimulation effects in disorders of consciousness. Arch Phys Med Rehabil. 2014 Feb;95(2):283-9. doi: 10.1016/j.apmr.2013.09.002. Epub 2013 Sep 11. PMID 24035769
- [Background] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549
- [Background] Thibaut A, Wannez S, Donneau AF, Chatelle C, Gosseries O, Bruno MA, Laureys S. Controlled clinical trial of repeated prefrontal tDCS in patients with chronic minimally conscious state. Brain Inj. 2017;31(4):466-474. doi: 10.1080/02699052.2016.1274776. Epub 2017 Mar 10. PMID 28281845
- [Background] Martens G, Lejeune N, O'Brien AT, Fregni F, Martial C, Wannez S, Laureys S, Thibaut A. Randomized controlled trial of home-based 4-week tDCS in chronic minimally conscious state. Brain Stimul. 2018 Sep-Oct;11(5):982-990. doi: 10.1016/j.brs.2018.04.021. Epub 2018 May 2. PMID 29759943
- [Background] Giacino JT, Kalmar K. Diagnostic and prognostic guidelines for the vegetative and minimally conscious states. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):166-74. doi: 10.1080/09602010443000498. PMID 16350959
- [Background] Sitt JD, King JR, El Karoui I, Rohaut B, Faugeras F, Gramfort A, Cohen L, Sigman M, Dehaene S, Naccache L. Large scale screening of neural signatures of consciousness in patients in a vegetative or minimally conscious state. Brain. 2014 Aug;137(Pt 8):2258-70. doi: 10.1093/brain/awu141. Epub 2014 Jun 11. PMID 24919971
- [Background] Engemann DA, Raimondo F, King JR, Rohaut B, Louppe G, Faugeras F, Annen J, Cassol H, Gosseries O, Fernandez-Slezak D, Laureys S, Naccache L, Dehaene S, Sitt JD. Robust EEG-based cross-site and cross-protocol classification of states of consciousness. Brain. 2018 Nov 1;141(11):3179-3192. doi: 10.1093/brain/awy251. PMID 30285102
- [Background] Bekinschtein TA, Dehaene S, Rohaut B, Tadel F, Cohen L, Naccache L. Neural signature of the conscious processing of auditory regularities. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1672-7. doi: 10.1073/pnas.0809667106. Epub 2009 Jan 21. PMID 19164526
- [Background] Faugeras F, Rohaut B, Weiss N, Bekinschtein T, Galanaud D, Puybasset L, Bolgert F, Sergent C, Cohen L, Dehaene S, Naccache L. Event related potentials elicited by violations of auditory regularities in patients with impaired consciousness. Neuropsychologia. 2012 Feb;50(3):403-18. doi: 10.1016/j.neuropsychologia.2011.12.015. Epub 2012 Jan 3. PMID 22230230